CLINICAL TRIAL: NCT05406635
Title: A National Randomized Non-inferiority Trial: Imaging Versus Cardiac Biomarker Monitored HER2 Directed Therapy in Patients With Breast Cancer
Brief Title: Imaging Versus Cardiac Biomarker Monitored HER2 Directed Therapy in Patients With Breast Cancer
Acronym: HER2BIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Collaborators: Aarhus University Hospital (Other); Aalborg University Hospital (Other); University of Copenhagen (Other)
Responsible Party: Principal Investigator, Ann Banke, Principal Investigator, Medical Doctor, PHD, Odense University Hospital
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OP_1413
Record Dates: First submitted 2022-05-12; First posted 2022-06-06 (Actual); Last update posted 2025-04-08 (Actual); Status verified 2025-04

CONDITIONS: Cardiotoxicity; HER2-positive Breast Cancer
MeSH Terms: conditions — Cardiotoxicity

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard imaging monitored treatment (No Intervention): Standard care + biomarkers, which are blinded until end of study.
- Intervention biomarker monitored treatment (Experimental): biomarker monitored treatment + imaging, which is blinded until end of study
  Interventions: Diagnostic Test: Biomarkers: Troponins and natriuretic peptides

INTERVENTIONS:
Diagnostic Test: Biomarkers: Troponins and natriuretic peptides — Biomarker monitored treatment with measurement of NT-proBNP and cTNT / TNI in weeks 0, 9, 18, 30 and 48 of the treatment period.
  Arms: Intervention biomarker monitored treatment

SUMMARY:
Due to a risk of heart failure during HER2 directed therapy in breast cancer, treatment is monitored with imaging of myocardial function, which is resource demanding for both patients and the health care system. The purpose of this study is to evaluate, if biomarkers can replace imaging based examinations of myocardial function during HER2 directed therapy.

DETAILED DESCRIPTION:
About 15% of breast cancer tumors express the Human Epidermal Growth Factor Receptor 2 (HER2), which is associated with a poor prognosis. Antibodies (trastuzumab and pertuzumab) directed against HER2 have in addition to traditional chemotherapy significantly improved survival in HER2 positive breast cancer, but induce a risk of left ventricular dysfunction and heart failure. Regular imaging based evaluation of myocardial function is therefore recommended during HER2 directed therapy by either an echocardiography or a MUGA scan, which is associated with radiation exposure. Both types of scans are resources demanding for both patients and the healthcare system, and since biomarkers have been proposed as another modality in assessment of myocardial injury, the purpose of this study is to evaluate, if biomarkers can replace imaging based examinations of myocardial function during HER2 directed therapy.

The study is designed as a national multicenter, randomized study, which will include Odense University Hospital, Herlev and Gentofte University Hospital and Aarhus University Hospital. It will be possible to include more sites.

Patients with localized HER2-positive breast cancer scheduled for HER2 proper therapy will be randomized 1: 1 to:

1. Standard imaging monitored treatment as recommended by DBCG guidelines with measurement of LVEF by MUGA scan or echocardiography in weeks 0, 9, 18, 30 and 48 of the treatment period. At each control visit, biomarkers are also taken, which are blinded until the end of the study.
2. Biomarker monitored treatment with measurement of NT-proBNP and cTNT / TNI in weeks 0, 9, 18, 30 and 48 of the treatment period. At each of these follow-up visits, MUGA scans or echocardiography are also performed, but the results are blinded to the staff responsible for treatment decisions.

In the group followed by standard imaging monitoring, cardiotoxicity will be managed according to standard clinical guidelines. Cardiotoxicity in the biomarker group will be suspected in case of a doubling of NT-proBNP from baseline (but minimum 125 pg / ml) and / or an increase in troponins to above 99th percentile. If these criteria are met, imaging is triggered, which in practice is a blinding of the result of the examination already performed.

The primary endpoint of the study is LVEF measured by cardiac MRI scan three months after completion of HER2-directed therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patients with non-metastatic HER2 positive breast cancer
* Scheduled for standard chemotherapy and HER2 directed therapy with trastuzumab +/- pertuzumab
* Age > 18 years
* Sinus rhythm on ECG
* NT-proBNP below125 pg/ml
* Troponin below threshold limit value
* LVEF > 55% by MUGA scan or an echocardiogram

Exclusion Criteria:

* Contra indications for cardiac magnetic resonance imaging (CMRI)
* Chronic obstructive pulmonary disease with FEV1 <80 % of predicted

Ages: 18 Years to 90 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 220 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2027-09-01 (Estimated)

PRIMARY OUTCOMES:
Left ventricular ejection fraction (LVEF) | Three months after treatment has ended.
  LVEF on cardiac MR.

SECONDARY OUTCOMES:
The number of treatment interruptions due to suspected cardiotoxicity | Through study completion, an average of 1 year.
  Number of times treatment was paused due to suspected cardiotoxicity either based on imaging or biomarkes as defined in the protocol.
The number of MUGA scans/echocardiograms | Through study completion, an average of 1 year.
  The number of MUGA scans/echocardiograms preformed during the study periode.
The cumulative doses of trastuzumab and pertuzumab | After end of treatment, an average of 1 year after inclusion.
  The cumulative doses of trastuzumab and pertuzumab in mg.
The proportion of patients treated for cardiotoxicity. | Through study completion, an average of 1 year
  Number of patients referred to tratment for heart failure in the department of cardiology.
Change in self-reported health status measured with EQ-5D-5L questionnaire | At baseline, at treatment week 9, 18, 30 and 48 and three months after end of treatment.
  An Index score and a Visual Analogue Scale (VAS).
Correlation between radiotherapy and cardiac function. | Through study completion, an average of 1 year
  Correlation between location and dose of the radiotherapy with changes in biomarkers, LVEF and ECG.

OTHER OUTCOMES:
Safty outcome of left ventricular ejection fraction | End of treatment
  Drop in LVEF below 45 %

CONTACTS AND LOCATIONS:
Overall Officials: Ann Banke, MD PHD, Principal Investigator — Odense Universitetshospital
Locations (4):
- Denmark (4):
  - Aalborg University Hospital, Aalborg
  - Rigshospitalet, Copenhagen
  - Herlev University Hospital, Herlev
  - Odense University Hospital, Odense

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- See also: Link to study description af Open Patient data Explorative Network — https://open.rsyd.dk/OpenProjects/openProject.jsp?openNo=1413&lang=da